CLINICAL TRIAL: NCT02641886
Title: A Study to Evaluate the Safety and Efficacy of Jian Pi Yi Shen Hua Tan Granules in Patients With Cognitive Impairment After Acute Cerebral Infarction
Brief Title: The Study of Jian Pi Yi Shen Hua Tan Granules in Cognitive Impairment After Acute Cerebral Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Collaborators: Changchun University of Chinese Medicine (Other); Chongqing Traditional Chinese Medicine Hospital (Other); Jiangmen Wuyi Hospital of Traditional Chinese Medicine (Other); Shunyi Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Yunling Zhang, President of Dongfang Hospital, Dongfang Hospital Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20140700108a
Record Dates: First submitted 2015-12-13; First posted 2015-12-30 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Impairment
Keywords: traditional Chinese medicine granules; Cognitive Impairment; Acute cerebral infraction; prevention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jian Pi Yi Shen Hua Tan Granules group (Experimental): Treat with the prescription of Jianpi Yishen Huatan Granules and conventional treatment of ischemic stroke.
  Interventions: Drug: Jian Pi Yi Shen Hua Tan Granules
- the Placebo Group (Placebo Comparator): Treat with the placebo which contain 5% of prescription of Jian Pi Yi Shen Hua Tan Granules and 95% dextrin and conventional treatment of ischemic stroke.
  Interventions: Other: the placebo group

INTERVENTIONS:
Drug: Jian Pi Yi Shen Hua Tan Granules — Jianpi Yishen Huatan Granules contain Herba cistanche，Fructus Alpinia Oxyphyllae，Rhodiola rosea, Polygala tenuifolia willd and Coptis chinensis.Jianpi Yishen Huatan Granules dissolved in water of 100 ml ,po, bid of each 90-days cycle. Number of treatment cycles: one
  Other Names: Jianpi Yishen Huatan Granules group
  Arms: Jian Pi Yi Shen Hua Tan Granules group
Other: the placebo group — Treat with the placebo which contain 5% of prescription of Jian Pi Yi Shen Hua Tan Granules and 95% dextrin.The placebo dissolved in water of 100 ml ,po, bid of each 90-days cycle. Number of cycles: one
  Arms: the Placebo Group

SUMMARY:
The purpose of this study is to determine whether the chinese medicine Jian Pi Yi Shen Hua Tan granules is effective in the treatment of cognitive impairment after acute cerebral infarction .

DETAILED DESCRIPTION:
The present study is designed to observe the symptoms,syndrome characteristics and neuropsychological changes of patients with cognitive dysfunction after Acute Cerebral Infarction, as well as study the patterns of syndrome evolution and neuropsychological characteristics, in order to provide evidences for the early-stage identification, diagnosis, intervention and treatment based on syndrome differentiation.

To assess the effectiveness of applying early-stage prevention on patients with cognitive impairment after Acute Cerebral Infarction through the use of traditional Chinese medicine--Jian Pi Yi Shen Hua Tan granules, explore the pathogenesis and therapeutic efficacy mechanism, evaluate the effectiveness of early-stage prevention and provide alternative solutions for preventing or delaying dementia.

ELIGIBILITY:
Inclusion Criteria:

* Patients conform to the diagnostic criteria of acute ischemic stroke Online Certificate Status Protocol classification of cerebral infarction : Partial Anterior Circulation Infarct, Posterior Circulation Infarct or Lacunar Infarction - Stroke onset within 14 days
* Neuropsychological assessments: Montreal Cognitive Assessment Scale scores less than 26 points or scores less than 27 points，MMSE scores range from 19 points to 26 points
* Age from forty to eighty, gender not limited
* Informed and signed the informed consent

Exclusion Criteria:

* Transient Ischemic Attack
* Online Certificate Status Protocol classification of cerebral infarction is a total anterior circulation infarction
* Stroke patients with the causes of cerebral hemorrhage, subarachnoid hemorrhage, brain tumors, brain injury, or blood diseases and so on.
* Stroke with an onset of more than 14 days
* Cerebral embolism caused by atrial fibrillation resulted from rheumatic heart disease, coronary heart disease and other heart diseases.
* Patients who cannot cooperate with the check due to serious visual, hearing dysfunction, apraxia, aphasia.
* Patients with other neurological diseases which can affect cognitive function (for example: severe Parkinson's disease, normal pressure hydrocephalus, brain tumors, encephalitis)
* Patients with communication difficulties, or psychiatric disease
* Depression (Hamilton Depression Scale scores more than or equal to 17 points) Diagnosed with alcohol or drug dependence within the past six months
* With other diseases which can cause cognitive dysfunction, Such as thyroid dysfunction, severe anemia, syphilis, Human Immunodeficiency Virus and so on
* With a previous history of stroke and serious sequelae, and cannot cope with neuropsychological examination
* With severe primary diseases, and cannot comply with the above scheme

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
mini-mental state examination | 90 days
  Using mini-mental state examination to examine the patients' cognitive function
Montreal Cognitive Assessment scale | 90 days
  Using Montreal Cognitive Assessment scale to examine the patients' cognitive function
Stroop test | 90 days
  Using Stroop test to examine executive function and attention
Numerical sequence test（DS-S) | 90 days
  Using Numerical sequence test（DS-S) to examine memeory
Digital color connection test (CCT) | 90 days
  Using Numerical sequence test（DS-S) to examine executive function and attention
Verbal memory test(HVLT) | 90 days
  Using Verbal memory test(HVLT) to examine verbal memory

SECONDARY OUTCOMES:
national institute of health stroke scale | 90 days
  Using national institute of health stroke scale to examine the neurologic function impairment
modified Rankin scale | 90 days
  Using modified Rankin scale to examine the recovery of neurologic function
Activity of Daily Living Scale | 90 days
  Using Activity of Daily Living Scale to examine daily living ability
scores of Chinese medicine symptoms | 90 days
  Using the scores of Chinese medicine symptoms to examine the Chinese medicine syndrom

CONTACTS AND LOCATIONS:
Overall Officials: Yunling Zhang, PhD,MD, Study Chair — Dongfang Hospital Beijing University of Chinese Medicine
Locations (5):
- China (5):
  - Department of Neurology,Dongfang Hospital, Beijing, Beijing Municipality
  - Shunyi Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Chongqing Hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - Jiangmen Wuyi Hospital of Traditional Chinese Medicine, Jiangmen, Guangdong
  - the Affiliated Hospital to Changchun University of Chinese Medicine, Changchun, Jilin